CLINICAL TRIAL: NCT04249258
Title: The Effects of Dobutamine on the Cardiac Conduction System: Site-Specific Dose
Brief Title: Dobutamine on the Cardiac Conduction System
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-0934
Record Dates: First submitted 2020-01-21; First posted 2020-01-30 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Dobutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dobutamine (Experimental): Measurements of various conduction parameters will be taken at baseline as is standard protocol for an EPS. Dobutamine will then be administered at doses of 5mcg/kg/min, 10mcg/kg/min, 15mcg/kg/min and 20mcg/kg/min. At each of these dosages the same conduction parameters will be measured. A comparison will then be made between the conduction parameters at baseline and when the Dobutamine is administered.
  Interventions: Drug: Dobutamine

INTERVENTIONS:
Drug: Dobutamine — Dobutamine will then be administered at doses of 5mcg/kg/min, 10mcg/kg/min, 15mcg/kg/min and 20mcg/kg/min.

SUMMARY:
Our hypothesis is that Dobutamine will act in a similar fashion to Isoproterenol with respect to cardiac conduction. Our goal is to study the effects of Dobutamine on cardiac conduction and refractoriness during an Electrophysiology study (EPS). At the end of most EPS Isoproterenol is commonly administered in an effort to change the conduction properties of the heart. In our practice we have been using Dobutamine for this purpose for many years. Dobutamine has never been rigorously studied for this indication however. We designed this study to systematically study the effect of various doses of Dobutamine on the parameters of cardiac conduction and refractoriness that are commonly measured during an EPS. We are specifically looking to compare the effect that Dobutamine has on the sinus node with the effect it has on the atrioventricular node. Patients undergoing an EPS at Long Island Jewish Hospital will be recruited and consented. Measurements of various conduction parameters will be taken at baseline as is standard protocol for an EPS. Dobutamine will then be administered at doses of 5mcg/kg/min, 10mcg/kg/min, 15mcg/kg/min and 20mcg/kg/min. At each of these dosages the same conduction parameters will be measured. A comparison will then be made between the conduction parameters at baseline and when the Dobutamine is administered.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, ages 18-80
4. Patients must be diagnosed with a condition that necessitates an EPS. They must also be deemed to be in good enough medical health to be eligible to safely undergo an EPS. Medical eligibility will be determined by the Attending Electrophysiologist performing the EPS.
5. For females of reproductive potential a negative pregnancy tes

Exclusion Criteria:

Patients with a resting left ventricular outflow gradient > 30mmHg

Patients with severe aortic stenosis

Patients with prior sustained ventricular tachycardia or ventricular fibrillation

Patients who are not able to consent for themselves

Patients with a prior allergic reaction to Dobutamine or any of its compounds including sulfites

Pregnant patients

Patients receiving B-blockers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
The change in sinus cycle length and anterograde atrioventricular node Wenckebach cycle length with Dobutamine | The sinus cycle length and anterograde AV node Wenckebach cycle length will be measured from baseline and at the end of 5 minutes of each dobutamine dose of 5mcg/kg/min, 10mcg/kg/min, 15mcg/kg/min and 20mcg/kg/min for a total of 20 minutes.
  The difference between the change in the sinus cycle length from baseline to the highest dose of Dobutamine compared to the change in the anterograde AV node Wenckebach cycle length from baseline to the highest dose of Dobutamine.

SECONDARY OUTCOMES:
The change in intervals measured in an EP study with Dobutamine | The parameters noted above will be measured at baseline and at the end of 5 minutes of each dose of dobutamine at 5mcg/kg/min, 10mcg/kg/min, 15mcg/kg/min and 20mcg/kg/min for a total of 20 minutes.
  The relative changes in baseline of escalating doses of Dobutamine on the sinus cycle length (msec), AH interval (msec), HV interval (msec), QRS duration (msec), QTc (msec), AV node Wenckebach cycle length (msec), AV node effective refractory period (msec) and VA block cycle length (msec).
The change in blood pressure with Dobutamine | The blood pressure will be measured at baseline and at the end of 5 minutes of each dose of dobutamine at 5mcg/kg/min, 10mcg/kg/min, 15mcg/kg/min and 20mcg/kg/min for a total of 20 minutes.
  The relative changes in baseline of escalating doses of Dobutamine on the blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Goldner, MD, Principal Investigator — Northwell Health
Locations (1):
- Long Island Jewish Hospital, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided